CLINICAL TRIAL: NCT07093424
Title: The Relationship of Magnesium Depletion Score With the Development of Complex Regional Pain Syndrome in Patients With Traumatic Extremity Injury
Brief Title: Relationship Between Complex Regional Pain Syndrome and Magnesium Depletion Score
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Dilara Ekici Zincirci, MD, Specialist, principal investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: RSD1
Record Dates: First submitted 2025-06-30; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-03

CONDITIONS: Complex Regional Pain Syndrome (CRPS)
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- traumatic extremity injury
  Interventions: Other: scoring

INTERVENTIONS:
Other: scoring — magnesium depletion score calculation

SUMMARY:
Complex Regional Pain Syndrome (CRPS) is a condition triggered by trauma such as surgery or a fracture. It is characterised by pain and limited mobility that are disproportionate to the severity of the trauma and the clinical course. Magnesium is recognised for its anti-inflammatory and antioxidant properties. The magnesium depletion score (MDS) is a more reliable and comprehensive scoring tool than measuring serum and urine magnesium levels. This score takes into account the patient's use of diuretics and proton pump inhibitors, their alcohol consumption, and their glomerular filtration rate. Impaired magnesium distribution may be a risk factor for CRPS development due to increased nociceptor activity. This study aimed to investigate whether an increased MDS score is a risk factor for CRPS development in individuals with traumatic limb injury.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-99 years with traumatic extremity injuries

Exclusion Criteria:

* History of previous stroke, spinal cord injury
* Presence of radiculopathy, radicular pain in the affected extremity
* Previous surgery for cervical discopathy/lumbar discopathy
* Presence of oncological, haematological diseases
* History of previous peripheral nerve injury or previous surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to our hospital's physical therapy and rehabilitation outpatient clinics with traumatic extremity injuries
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
CRPS development | baseline
  crps development will be assessed according to Budapest criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu Şehir Hastanesi, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF